CLINICAL TRIAL: NCT01274949
Title: The Effect of Low Intensity Shock Wave Therapy in Post Radical Prostatectomy Severe ED Patients Not Responding to Oral Medication
Brief Title: The Effect of Low Intensity Shockwave Therapy for ED in Post Radical Prostatectomy Patients Who Didn't Respond to PDE5i
Acronym: LI-ESWT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Medispec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3060 radical
Record Dates: First submitted 2011-01-09; First posted 2011-01-12 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Erectile Dysfunction
Keywords: LI-ESWT; Erectile Dysfunction; Radical Prostatectomy; Non PDE5 inhibitor responders; Shock wave
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LI-ESWT (Experimental): Low intensity shock wave treatment- 12 sessions
  Interventions: Device: LI-ESWT

INTERVENTIONS:
Device: LI-ESWT — Low intensity shock wave treatment - 12 sessions
  Other Names: Omnispec model ED1000

SUMMARY:
Low Intensity Shock Wave Therapy (LI-ESWT) was shown to have a beneficial effect on ED patients responding to PDE5i's. This study aimed to determine the capability of LI-ESWT to affect patients who underwent radical prostatectomy who did not respond to PDE5 inhibitor therapy.

DETAILED DESCRIPTION:
We included severe ED patients that underwent radical prostatectomy at least one year previously and failed to respond to PDE5i therapy, who scored 0-2 on the rigidity scale (RS) during PDE5i therapy. Treatment included 2 sessions/week for 3 weeks, repeated after a 3-week no-treatment interval. At each session LI-ESWT was applied on the penile shaft and crus for 3 minutes in 5 different penile anatomical sites (intensity of 0.09 mj/mm2, 300 shocks/site). One-month after end of treatment the same baseline assessment was repeated. An active PDE5i medication regime was then provided and final erectile function was reassessed. Main endpoints for success were changes in RS and in the International Index of Erectile Function (IIEF-ED) Domain score. This study further emphasises the need to study specific populations with unique etiologies causing ED.

ELIGIBILITY:
Inclusion Criteria:

* Post Radical prostatectomy
* ED of more than 6 months
* Rigidity score ≤ 2 during PDE5i therapy
* Stable heterosexual relationship for more than 3 months
* Patients need to know and to agree that the study protocol does not allow any PDE5I therapy till week 13 .

Exclusion Criteria:

* Prior surgery or radiotherapy in pelvic region
* Any unstable, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Cardiovascular conditions that prevent sexual activity

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
IIEF-ED Domain score | 17 weeks after first visit
  Change of 5 points and above in IIEF-ED Domain score

SECONDARY OUTCOMES:
Rigidity scale | 17 weeks after first visit
  a change to 3 or 4 points in the rigidty scale

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Study Director — Rambam Medical Investigator
Locations (1):
- neuro-urology unit, Rambam Medical Center, Haifa, Israel